CLINICAL TRIAL: NCT03592459
Title: Rectal Administration of Opioids for Comfort Care in Advanced Cancer Patients Using the Macy Catheter
Brief Title: Rectal Administration of Opioids Using the Macy Catheter in Reducing Pain in Patients With Advanced Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-0321; NCI-2018-01344 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0321 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Advanced Malignant Neoplasm; Pain
MeSH Terms: conditions — Pain | interventions — Analgesia; Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device feasibility (Macy catheter, opioids) (Experimental): Patients undergo placement of rectal catheter and receive opioids through the Macy catheter.
  Interventions: Device: Macy Catheter; Procedure: Pain Therapy; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Device: Macy Catheter — Undergo placement of Macy catheter
Procedure: Pain Therapy — Receive opioids via Macy catheter
  Other Names: analgesia; Pain Control; Pain Management; Pain, Pain Management
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well rectal administration of opioids using the Macy catheter works in reducing pain in patients with cancer that has spread to other anatomic sites or is no longer responding to treatment. Rectal administration of opioids using the Macy catheter may help to reduce the cost of care, resolve the issue of medication availability currently faced in the form of parenteral opioid shortage throughout the country, and provide adequate comfort and symptom relief for patients with smoother transition out of hospital.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of using the device 'Macy catheter' for rectal administration of opioids for comfort in cancer patients on palliative care.

SECONDARY OBJECTIVES:

I. To determine the ease of use, level of satisfaction and overall perception of effectiveness of 'Macy catheter' for rectal administration of opioids for pain control in advanced cancer patients, by the hospital bedside nursing staff.

II. To assess patients' (or primary care-giver's) experience of using the 'Macy catheter' 48 hours after discharge from the hospital.

III. To assess the hospice staff (or primary care-giver's) experience of using the 'Macy catheter' after patient's death.

OUTLINE:

Patients undergo placement of rectal catheter and receive opioids through the Macy catheter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the inpatient Acute Palliative Care Unit (APCU) at MD Anderson Cancer Center
* Candidate for taking short acting opioids and/or methadone, with or without transdermal fentanyl, for control of cancer related pain
* Impaired oral/gastrointestinal (GI) route for medicine intake (due to, but not limited to, any level of gastrointestinal obstruction, severe nausea and/or vomiting, odynophagia and/or dysphagia due to severe mucositis, tumor, muscle weakness or in-coordination)
* Advanced cancer defined as cancer with no further oncological management and patients are at end of life (EOL) or recommended for best supportive/comfort care (estimated prognosis less than 6 months)
* Able and willing to read and sign in English

Exclusion Criteria:

* Non-English speaking
* Contraindications to use of the Macy catheter (1. Not be used for patients with rectal lesions, tumors, active rectal bleeding and/or compromised rectal mucosa [i.e. ulceration or ischemic proctitis], 2. Patients with diarrhea, or more than 1 liquid stool per day, 3. Patients with recent bowel surgery [less than 6 weeks], 4. Thrombocytopenia [platelet count less than 20,000, checked in the last 1 week])
* Patients who are unable to take oral medications due to severe constipation only, which can be adequately managed by bowel laxative regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the device 'Macy catheter' for rectal administration of opioids for comfort in cancer patients on palliative care as defined by number of doses administered and patient satisfaction | Up to 1 year
  Will be assessed by the number of doses that a patient finishes (at least 4 out of 6 doses administered) and by asking patients' about their level of satisfaction and overall perception of effectiveness of using the device, collected by question 10 and 11 in the survey, respectively. The association between patients' demographics and clinical characteristics and patients' satisfaction and perception of effectiveness will be evaluated by Wilcoxon rank sum test and chi-square (or Fisher's exact) test for continuous and categorical variables, respectively. In order to address the primary objective, the feasibility rate will be estimated and reported along with a 95% Clopper-Pearson exact confidence interval.

SECONDARY OUTCOMES:
Episodes of confusion (delirium) assessed by primary caregiver survey | Up to 1 year
Hospice nurse experience assessed by survey | Up to 1 year
  Will be summarized by frequency tables. McNemar's test will be applied to evaluate whether the feasibility changes from the time at the hospital to 48 hours of discharge. Other statistical methods may be applied when appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Azhar, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org